CLINICAL TRIAL: NCT05050903
Title: Early Antiviral Responses to Rhinovirus Infection in Asthma
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21SM6879
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma
  Interventions: Other: Rhinovirus infection
- Healthy controls
  Interventions: Other: Rhinovirus infection

INTERVENTIONS:
Other: Rhinovirus infection — Inoculation with rhinovirus-16

SUMMARY:
The bulk of the morbidity and mortality related to asthma is during periods of acutely increased symptomatology called 'exacerbations'. Roughly half of asthma sufferers experience such an exacerbation each year. Most of these events are triggered by viral infections, usually the common cold virus (rhinovirus).

A key part of the body's defence against viral infections is to produce antiviral proteins called 'interferons', which have a myriad of effects to stop viruses. Previous work on cells taken from volunteers with asthma and healthy controls and infected with rhinovirus in the lab suggests interferon production is impaired in asthma. However when human volunteers with asthma are infected with rhinovirus, high levels of interferon are found a few days later - along with high numbers of virus. Whether the high virus numbers are the result of an initially weak interferon response, with subsequently unchecked viral replication leading to exaggerated interferon levels, is unknown as no one has measured interferons early in infection.

By infecting volunteers with asthma and healthy controls with rhinovirus at a known time, only done in a handful of centres worldwide, we will be able to measure interferons within hours of infection and well before symptoms develop.

ELIGIBILITY:
For Asthma group:

Inclusion Criteria:

* Age 18-55 years
* Doctor diagnosis of asthma
* Previous asthma exacerbation

Exclusion Criteria:

* Smoking history over past 12 months
* Sinonasal disease, including current symptoms of allergic rhinitis
* Asthma exacerbation or an upper respiratory viral infection within the previous six weeks
* Current or concomitant use of oral steroids, monoclonal antibodies or nasal sprays
* Neutralising antibodies to rhinovirus (RV)-16
* Clinically significant diseases other than asthma which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, influence the results of the study, an/or the patient's ability to take part in it
* Inability to understand written or verbal information in English

For healthy control group:

Inclusion Criteria:

• Age 18-55 years

Exclusion Criteria:

As for Asthma group and in addition:

• History of asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Potential participants will be identified from hospital outpatient clinics, primary care, spirometry sessions/clinics, other research projects, and advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Nasal IFN-λ at 6 hours post rhinovirus infection | 6 hours
  Difference in IFN-λ in nasal lining fluid 6 hours following rhinovirus infection in subjects with asthma compared to healthy controls

SECONDARY OUTCOMES:
Nasal IFN-α at 6 hours post rhinovirus infection | 6 hours
  Difference in IFN-α in nasal lining fluid 6 hours following rhinovirus infection in subjects with asthma compared to healthy controls
Nasal IFN-λ at 3 hours post rhinovirus infection | 3 hours
  Difference in IFN-λ in nasal lining fluid 3 hours following rhinovirus infection in subjects with asthma compared to healthy controls
Nasal IFN-λ at 24 hours post rhinovirus | 24 hours
  Difference in IFN-λ in nasal lining fluid 24 hours following rhinovirus infection in subjects with asthma compared to healthy controls
Nasal IFN-α at 3 hours post rhinovirus infection | 3 hours
  Difference in IFN-α in nasal lining fluid 3 hours following rhinovirus infection in subjects with asthma compared to healthy controls
Nasal IFN-α at 24 hours post rhinovirus infection | 24 hours
  Difference in IFN-α in nasal lining fluid 24 hours following rhinovirus infection in subjects with asthma compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Johnston, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Respiratory Research Unit, St Mary's Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No